CLINICAL TRIAL: NCT05017168
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Parallel Group, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of CT-P63 in Healthy Subjects
Brief Title: To Evaluate the Safety, Tolerability and Pharmacokinetics of CT-P63 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P63 1.1; 2021-003530-37 (EudraCT Number)
Record Dates: First submitted 2021-07-29; First posted 2021-08-23 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — CT-P63

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-P63 (Experimental): Single Ascending Dose
  Interventions: Drug: CT-P63
- Placebo (Placebo Comparator): Single Ascending Dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT-P63 — CT-P63 will be administered
  Arms: CT-P63
Drug: Placebo — Placebo-matching CT-P63
  Arms: Placebo

SUMMARY:
This is a Phase I study that randomized, double-blind, Placebo-controlled, Parallel Group, Single Ascending Dose Study to evaluate Safety, Tolerability and Pharmacokinetics of CT-P63 in Healthy Subjects.

DETAILED DESCRIPTION:
CT-P63 is a monoclonal antibody targeted against SARS-CoV-2 spike RBD as a treatment for SARS CoV 2 infection. CT-P63 is currently being developed by the Sponsor as a potential treatment for SARS-CoV-2 infection. In this study, safety, tolerability, and pharmacokinetics of CT-P63 will be evaluated in healthy subjects.

ELIGIBILITY:
[Inclusion Criteria]

Each subject must meet all of the following criteria to be randomized in this study:

1. Subject is a healthy male or female subject, aged between 18 to 60 years (both inclusive). Health is defined as no clinically relevant abnormalities identified by Investigator's decision based on a detailed medical history, full physical examination, including blood pressure, heart rate, respiratory rate, and body temperature measurements, 12-lead electrocardiogram (ECG) and clinical laboratory tests prior to the study drug administration.
2. Subject with a body weight of ≥ 50 kg and a body mass index between 18.0 and 29.9 kg/m2 (both inclusive).
3. Subject is able to understand and to comply with protocol requirements, instructions, and restrictions.

[Exclusion Criteria]

A Subject meeting any of the following criteria will be excluded from the study:

1. Subject has a medical history or current presence of disease including one or more of the following(s):

   1. History of or current allergic reaction such as asthma, urticaria, angioedema, and eczematous dermatitis considered as clinically significant in the Investigator's opinion or hypersensitivity including known or suspected clinically relevant drug hypersensitivity to any monoclonal antibody or any component of study drug
   2. History of or current medical condition including gastrointestinal, renal, endocrine, neurologic, autoimmune, hepatic, hematological metabolic (including known diabetes mellitus), cardiovascular, or psychiatric condition classed as clinically significant by the Investigator
   3. History of malignancy within past 5 years or any current malignancy
   4. Current infection with human immunodeficiency, syphilis, hepatitis B or hepatitis C
   5. History of or current infection requiring a course of systemic anti-infective that was completed within 28 days prior to the study drug administration or a serious infection (associated with hospitalization or which required IV antibiotics) within 6 months before the study drug administration
   6. History of an illness within 28 days prior to the study drug administration that is identified as clinically significant by the Investigator or requires hospitalization
   7. History of surgical intervention or an operation within 28 days prior to the study drug administration or plans to have a surgical procedure during the study period
2. Subject had a history of or concurrent use of medications including any prior therapy of following(s):

   1. Any vaccination within 4 weeks prior to the study drug administration. For SARS-CoV-2 vaccine, subject who received any investigational or approved SARS-CoV-2 vaccine cannot be enrolled, regardless of the timing of administration
   2. Treatment with any monoclonal antibody, fusion protein, or blood transfusion within 6 months or 5 half lives (which is longer) prior to the study drug administration or current use of biologics
   3. Prescription medication (excluding hormonal birth control), over-the-counter drug, dietary supplements or herbal remedies within 7 days or 5 half-lives (whichever is longer) prior to the study drug administration
   4. Treatment with any other investigational drug within 6 months or 5 half lives (which is longer) prior to the study drug administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of single ascending dose of CT-P63: | Up to 14 Days
  1. Proportion of patients with Treatment Emergent Adverse Events (TEAEs) by CTCAE v5.0
  2. Proportion of patients with Treatment Emergent Serious Adverse Events (TESAEs) by CTCAE v5.0
  3. Proportion of patients with TEAEs of special interest (IRR including hypersensitivity/anaphylactic reaction) by CTCAE v5.0

SECONDARY OUTCOMES:
To evaluate immunogenicity of single ascending dose of CT-P63: | Up to 90 Days
  Incidence of ADA and NAbs to CT-P63 (positive or negative)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  Pharmacokinetic (PK) parameter: Area under the serum concentration-time curve from time zero to infinity, calculated using the linear up and low down trapezoidal rule(AUC0-inf)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Dose normalized AUC0-inf (normalized to total body dose)(AUC0-inf/Dose)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Area under the serum concentration-time curve from time zero to the last quantifiable concentration, calculated using the linear up and log down trapezoidal rule(AUC0-last)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Dose normalized AUC0-last (normalized to total body dose)(AUC0-last/Dose)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Maximum observed serum concentration(Cmax)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Dose normalized Cmax(normalized to total body dose)(Cmax/Dose)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Time to Cmax(Tmax)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Terminal elimination half-life(t1/2)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Percentage of the area extrapolated for calculation of AUC0-inf(%AUCext)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Terminal elimination rate constant estimated from the linear regression of the natural log-transformed concentration over time at the terminal phase(λz)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Total body clearance(CL)
To evaluate the Pharmacokinetic(PK) of CT-P63 | Up to 90 Days
  PK parameter: Volume of distribution at steady state (Vss)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Kiecana, Dr., Principal Investigator — Biokinetica S.A.
Locations (1):
- Biokinetica S.A, Józefów, Poland